CLINICAL TRIAL: NCT00030810
Title: Preoperative Chemoradiotherapy In Non-Small Cell Lung Cancer (NSCLC) Patients With Operable Stage IIIB Disease: A Prospective Phase II Trial
Brief Title: Combination Chemotherapy Followed by Radiation Therapy Before Surgery in Treating Patients With Stage IIIB NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 16/01; EU-20137
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Hyperfractionated — Hyperfractionated radiotherapy
Drug: Taxotere/Cisplatin — Taxotere/Cisplatin
Procedure: conventional surgery — conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by radiation therapy before surgery in treating patients who have stage IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and efficacy of sequential neoadjuvant docetaxel, cisplatin, and radiotherapy followed by surgery in patients with operable stage IIIB non-small cell lung cancer.
* Determine the rate of event-free survival at 1 year in patients treated with this regimen.
* Determine the operability and complete resection rate in patients treated with this regimen.
* Determine the postoperative 30-day mortality in patients treated with this regimen.
* Determine the response rate, failure pattern, and overall survival in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of unacceptable toxicity.

Beginning 3 weeks after the last chemotherapy dose, patients without progressive disease receive radiotherapy 1-2 times daily on days 1-5, 8-12, and 15-19.

Patients undergo surgery within 3-4 weeks after completion of radiotherapy.

Patients are followed at 1 month and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 15-46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, operable stage IIIB non-small cell lung cancer

  * T4 N0-3 M0 or T1-4 N3 M0 by bronchoscopy and mediastinoscopy (required for assessment of N3 disease) or CT scan or MRI of the thorax
  * Squamous cell
  * Adenosquamous cell
  * Large cell
  * Poorly differentiated
* No prior or concurrent metastatic disease by CT scan or MRI of the brain, bone scan, and abdominal ultrasound or CT scan
* No malignant pleural or pericardial effusion
* No invasion of the aorta, esophagus, myocardium, or supraclavicular nodes

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST and/or ALT no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No unstable cardiac disease requiring treatment
* No congestive heart failure
* No angina pectoris (even if medically controlled)
* No significant arrhythmia
* No myocardial infarction within the past 3 months

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No definite contraindications for the use of corticosteroids as premedication
* No preexisting grade 2 or greater peripheral neuropathy
* No active uncontrolled infection
* No uncontrolled diabetes mellitus
* No other prior or concurrent malignancy except non-melanomatous skin cancer or adequately treated carcinoma in situ of the cervix
* No prior significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures that would preclude informed consent
* No other serious underlying medical condition that would preclude study participation
* No socioeconomic or geographical circumstances that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent corticosteroids except as prophylactic pretreatment medication, treatment for acute hypersensitivity reactions, or chronic treatment (initiated more than 6 months ago) at low-dose (no more than 20 mg methylprednisolone or equivalent)

Radiotherapy:

* No prior radiotherapy to the chest

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since prior treatment in a clinical trial
* No prior cytostatic therapy
* No other concurrent experimental drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Rate of event-free survival measured 1 year after registration

SECONDARY OUTCOMES:
Operability after chemotherapy
Postoperative mortality 30 days after surgery
Complete resection rate after surgery
Toxicity
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Stupp R, Mayer M, Kann R, Weder W, Zouhair A, Betticher DC, Roth AD, Stahel RA, Majno SB, Peters S, Jost L, Furrer M, Thierstein S, Schmid RA, Hsu-Schmitz SF, Mirimanoff RO, Ris HB, Pless M. Neoadjuvant chemotherapy and radiotherapy followed by surgery in selected patients with stage IIIB non-small-cell lung cancer: a multicentre phase II trial. Lancet Oncol. 2009 Aug;10(8):785-93. doi: 10.1016/S1470-2045(09)70172-X. Epub 2009 Jul 13. PMID 19604722
- [Result] Pless M, Stupp R, Kann R, et al.: Preoperative chemoradiotherapy in non-small cell lung cancer (NSCLC) patients with operable stage IIIB disease: a phase II trial of the Swiss Group for Clinical Cancer Research (SAKK). [Abstract] J Clin Oncol 25 (Suppl 18): A-18021, 685s, 2007.
- [Result] Fruh M, Betticher DC, Stupp R, Xyrafas A, Peters S, Ris HB, Mirimanoff RO, Ochsenbein AF, Schmid R, Matzinger O, Stahel RA, Weder W, Guckenberger M, Rothschild SI, Lardinois D, Mach N, Mark M, Gautschi O, Thierstein S, Biaggi Rudolf C, Pless M; Swiss Group for Clinical Cancer Research (SAKK). Multimodal Treatment in Operable Stage III NSCLC: A Pooled Analysis on Long-Term Results of Three SAKK trials (SAKK 16/96, 16/00, and 16/01). J Thorac Oncol. 2019 Jan;14(1):115-123. doi: 10.1016/j.jtho.2018.09.011. Epub 2018 Sep 26. PMID 30267838
- [Result] Fruh M, Ris HB, Xyrafas A, Peters S, Mirimanoff RO, Gautschi O, Pless M, Stupp R. Preoperative chemoradiotherapy with cisplatin and docetaxel for stage IIIB non-small-cell lung cancer: 10-year follow-up of the SAKK 16/01 trial. Ann Oncol. 2016 Oct;27(10):1971-3. doi: 10.1093/annonc/mdw251. Epub 2016 Jun 29. No abstract available. PMID 27358380